CLINICAL TRIAL: NCT01729663
Title: Randomized, Comparative Phase II/III Study Between Treatment With CSF470 Vaccine (Allogeneic, Irradiated) Plus BCG and MOLGRAMOSTIN (rhGM-CSF) as Adjuvants and Interferon-alfa 2b (IFN-ALPHA), in Stages IIB, IIC and III Post Surgery Cutaneous Melanoma Patients
Brief Title: Phase II/III Clinical Study CSF470 Plus BCG Plus GM-CSF vs IFN Alpha 2b in Stage IIB, IIC and III Melanoma Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorio Pablo Cassará S.R.L. (Industry)
Collaborators: Fundacion Sales (Unknown); National Agency for Scientific and Technological Promotion, Argentina (Other); Fundacion Cancer FUCA (Unknown); National Council of Scientific and Technical Research, Argentina (Other Government); Instituto Nacional del Cáncer, Argentina (Other Government)
Responsible Party: Principal Investigator, José Mordoh, MD, PhD, Laboratorio Pablo Cassará S.R.L.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASVAC0401
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Cutaneous Melanoma
Keywords: melanoma; irradiated-allogeneic cells; therapeutic vaccine; Interferon alpha 2-b
MeSH Terms: conditions — Melanoma | interventions — molgramostim; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interferon alpha 2 b (Active Comparator): Interferon alpha 2b treatment will consist of s.c. injection of 10 MU (5 t/w) for four weeks and then 5 MU (3t/w) for 23 months.
  Interventions: Drug: interferon alpha 2b
- CSF470 vaccine, BCG, Molgramostim (Experimental): CSF470 vaccine, BCG, Molgramostim
  CSF-470 treatment will consist of four vaccine doses id injection (three weeks apart), then one dose every two months for the first year and them every three months for the second year.
  Each vaccine consist of a mixture of 17,6.106 melanoma cells , from four melanoma cell lines, not genetically modified and lethally irradiated. As adjuvant BCG (120 µg prot) the first day and rhGM-CSF (Molgramostim 400 µg, fractionated in four days doses) will be used.
  Interventions: Biological: CSF470 vaccine, BCG, Molgramostim

INTERVENTIONS:
Biological: CSF470 vaccine, BCG, Molgramostim
  Arms: CSF470 vaccine, BCG, Molgramostim
Drug: interferon alpha 2b
  Arms: Interferon alpha 2 b

SUMMARY:
Randomized, open, Phase II-III study, comparative between treatment with CSF-470 vaccine , allogeneic, irradiated with BCG and molgramostin (rHuGM-CSF) as adjuvants and interferon alfa 2b (IFN-alpha2b) treatment , in stages IIB, IIC o III (AJCC) post-surgery cutaneous melanoma patients. This study has been approved by ANMAT ( Administración Nacional de Medicamentos, Alimentos y Tecnología Médica (ANMAT)), number 1556/2011 (www.anmat.gov.ar).

The study Institution is Instituto Médico Especializado Alexander Fleming, Ciudad Autónoma de Buenos Aires, Argentina. The Sponsor is Laboratory Pablo Cassará (LPC, S.R.L.).

Study population include a total of 108 patients (72 patients will receive CSF470 vaccine and 36 patients will receive alpha IFN-alpha 2b) for a total of 24 months.

CSF-470 treatment will consist of four vaccine doses id injection (three weeks apart), then one dose every two months for the first year and them every three months for the second year.

Each vaccine consist of a mixture of 17,6.106 melanoma cells, from four melanoma cell lines, not genetically modified and lethally irradiated. As adjuvant BCG (120 µg prot) the first day and rHuGM-CSF (Molgramostim, 400 µg, fractionated in four days doses) will be used.

IFN-alpha 2b treatment will consist of s.c. injection of 10 million units (MU) (5 t/w ) for four weeks and then 5 MU (3t/w) for 23 months.

Both treatments will also compare quality of life (QOL) and study a possible correlation in the CSF470 vaccine arm between the induced immune response and clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed cutaneous melanoma stages IIB, IIC or III (AJCC)
* patients non-detectable disease (NED) after surgery as asserted by CAT scans. Melanoma pts with unknown primary tumor site could be included in the study
* life expectancy > 6 months
* performance status (ECOG) 0 or 1
* Time post surgery not more than 4 months
* no chemotherapy, radiotherapy or any biological treatments prior to this study.
* patients must have CATscans of brain, thorax, abdomen and pelvis in the 60 previous days to trial enrolling
* To have laboratory studies (no more than 15 days before entering the study)
* laboratory eligibility criteria include: hematocrit: ≥35 (hemoglobin > 10,5 gr %); WBC count > 3500/mm3, platelets > 100.000/mm3, total and direct bilirubin, serum oxalacetic transaminase and glutamic pyruvic transaminase < 1.5 fold the upper normal value; LDH ≤ 450 mU/ml
* negative serology for HIV, anti-HCV and HBsAg
* serum creatinine < 2.0 mg %
* all patients must give written informed consent before inclusion in the Study.

Exclusion Criteria:

* Pregnant or breast-feeding women
* Diabetes (Type I or II)
* Antecedents of psychiatric diseases
* Evidence of active infections
* Antecedents of viral or autoimmune hepatitis
* Previous autoimmune diseases
* Morbid Obesity, defined as CMI (Corporal mass index)>37 kg/m2 in women and >40 kg/m2 in men.
* Other diseases that require treatment with regular corticoids or non steroids anti-inflammatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2009-04; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy | two years
  OS, DFS, Partial or total remission (PR or CR)
security | two years
  measured according to the NCI-Common Toxicity Criteria

SECONDARY OUTCOMES:
Quality of Life | two years
  QOL:evaluated with EORTC QLQ-C30 questionnaire; ECOG Performance status
Induction of immune responses | two years
  Induction of immune responses associated to different vaccine doses for 2 years (Trial duration) ]Cellular immunity (DTH) - Humoral immunity

CONTACTS AND LOCATIONS:
Overall Officials: José Mordoh, MD, PhD, Principal Investigator — Instituto Médico Alexander Fleming
Locations (1):
- Instituto Médico Alexander Fleming, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Derived] Aris M, Bravo AI, Pampena MB, Blanco PA, Carri I, Koile D, Yankilevich P, Levy EM, Barrio MM, Mordoh J. Changes in the TCRbeta Repertoire and Tumor Immune Signature From a Cutaneous Melanoma Patient Immunized With the CSF-470 Vaccine: A Case Report. Front Immunol. 2018 May 3;9:955. doi: 10.3389/fimmu.2018.00955. eCollection 2018. PMID 29774030
- [Derived] Mordoh J, Pampena MB, Aris M, Blanco PA, Lombardo M, von Euw EM, Mac Keon S, Yepez Crow M, Bravo AI, O'Connor JM, Orlando AG, Ramello F, Levy EM, Barrio MM. Phase II Study of Adjuvant Immunotherapy with the CSF-470 Vaccine Plus Bacillus Calmette-Guerin Plus Recombinant Human Granulocyte Macrophage-Colony Stimulating Factor vs Medium-Dose Interferon Alpha 2B in Stages IIB, IIC, and III Cutaneous Melanoma Patients: A Single Institution, Randomized Study. Front Immunol. 2017 May 31;8:625. doi: 10.3389/fimmu.2017.00625. eCollection 2017. PMID 28620382